CLINICAL TRIAL: NCT01376947
Title: Comparison of the Difficulty on Insertion of IUD Devices Between Nulliparous and Multiparous and Evaluation of Cause of Failure of Insertion
Brief Title: Comparison of the Difficulty on Insertion of IUD Devices Between Nulliparous and Multiparous Women
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Center for Research on Reproductive Health of Campinas (Other)
Responsible Party: Ana Raquel Gouvea Santos, MAster degree student
Other Study IDs: 02/2011/PC
Record Dates: First submitted 2011-04-24; First posted 2011-06-20 (Estimated); Last update posted 2011-06-20 (Estimated); Status verified 2011-06

CONDITIONS: Complication of Device Insertion
Keywords: IUD device insertion; Nulliparous; Multiparous; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Nulliparous: Nulliparous women who were submitted to IUD device insertion
- Multiparous with no cesaraen section: Multiparous women with no cesarean sections that were submitted to IUD device insertion
- Mulitparous with cesarean section: multiparous women with a cesarean section that were submitted to IUD insertion

SUMMARY:
In this study the investigators compare the difficulty at insertion of IUD between nulliparous and parous women. The investigators compare the pain reported by the patient to the difficulty reported by the professional that performed the insertion.

The investigators hypothesis is that there is no difference between nulliparous and multiparous patients.

DETAILED DESCRIPTION:
In our study we compare the difficulty at insertion of IUD between nulliparous and parous women with an without cesarean section.

We compare the pain reported by the patient to the difficulty reported by the professional that performed the insertion. We also compare the pain the patient refers on the day of insertion and the pain the patient refers to remember a month after insertion.

Our hypothesis is that there is no difference between nulliparous and multiparous patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy WOmen

Exclusion Criteria:

* Pregnancy
* Use of pain medication previous to the insertion
* Prior use of IUDs

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy women that desire to use IUD as anticonceptional method
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-06 (Estimated); Study Completion 2011-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Raquel Gouvea Santos, MD, Principal Investigator — UNICAMP - master degree student; Ilza Urbano, PHD, Study Director — Professor at UNICAMP
Locations (1):
- UNICAMP - Departamento de Tocoginecologia, Campinas, São Paulo, Brazil